CLINICAL TRIAL: NCT07155343
Title: Comparison of the Brackets Bonded With Bulk Fill Composite and Conventional Composite in Patients Undergoing Fixed Orthodontic Treatment - A Split-mouth Randomized Controlled Trial
Brief Title: Comparison of the Brackets Bonded With Bulk Fill Composite and Conventional Composite in Patients Undergoing Fixed Orthodontic Treatment
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rizwan Khalil (Other)
Collaborators: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Sponsor-Investigator, Rizwan Khalil, Resident Orthodontic, Aga Khan University Hospital, Pakistan
Organization: Aga Khan University Hospital, Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-9142-30284
Record Dates: First submitted 2025-07-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Survival Rate of Bonded Brackets
Keywords: Bulk fill composite; Bond failure rate; Fixed orthodontic treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brackets Bonded Using Bulk Fill Composite (Experimental): In this arm, orthodontic brackets will be bonded using a light-cured bulk fill composite resin material. The composite will be applied directly to the bracket base and cured according to the manufacturer's instructions. This group is intended to evaluate the clinical performance, bond failure rate, and handling characteristics of bulk fill composite in comparison to conventional orthodontic bonding resin. Brackets will be placed on either the right or left side of the arch, based on random allocation.
  Interventions: Combination Product: Bulk Fill Composite
- Brackets Bonded Using Conventional Composite (Active Comparator): In this arm, orthodontic brackets will be bonded using a conventional light-cured orthodontic composite resin. The composite will be applied to the bracket base and cured according to the manufacturer's recommended protocol. This group will serve as the control to compare the bond strength, failure rate, and clinical performance against the bulk fill composite group. Brackets will be placed on either the right or left side of the arch, depending on the random allocation.
  Interventions: Combination Product: Conventional Composite

INTERVENTIONS:
Combination Product: Bulk Fill Composite — Orthodontic brackets will be bonded using a bulk fill composite resin, which is formulated for faster application and reduced polymerization shrinkage compared to conventional composites. This material will be used to assess its bond strength, failure rate, and overall clinical performance.
  Arms: Brackets Bonded Using Bulk Fill Composite
Combination Product: Conventional Composite — Orthodontic brackets will be bonded using a conventional light-cured orthodontic composite resin that requires careful incremental application and standard curing time. This material is commonly used in routine clinical practice and serves as the benchmark for comparison.
  Arms: Brackets Bonded Using Conventional Composite

SUMMARY:
The primary objective of this study is to compare the survival rate (days) of orthodontic bracket bond to the tooth, and the secondary objective is to compare the dental plaque accumulation and gingival health using plaque index and gingival index respectively between brackets bonded with bulk fill composite and light cure conventional composite in patients undergoing fixed orthodontic treatment over a period of three months.

DETAILED DESCRIPTION:
After obtaining approval from the Ethical Review Committee and taking informed assent and informed consent from the child and parents respectively, patients fulfilling the study selection criteria will be recruited in the study as participants. Patients visiting the orthodontic clinic at the Aga Khan University Hospital Karachi will be included in this study. Detailed information regarding the study will be provided to the participants and they will be given the choice to either accept or refuse their inclusion in the study. Bulk fill composite and light cure conventional composite will be used to bond the brackets in the study participants undergoing orthodontic treatment. Bulk fill composite and light cure conventional composite will be randomly allocated to the right and left quadrants of maxillary and mandibular arches. Bracket bond failure and clinical measurements (plaque accumulation and gingival health) will be recorded at four intervals. First, at the time of brackets bonding (T0), after one month (T1), two months (T2) and three months follwow-up (T3). Data will be collected on an organized study proforma.

Interim analysis will be run to ensure that there are no unexpected safety concerns associated with the intervention. The analysis may help determine whether the intervention is effective in achieving its desired outcomes or if there are indications of potential success. If the interim analysis will reveal overwhelming evidence of effectiveness or futility, the trial will be terminated early, saving time, money, and potential exposure to participants.

Intention to treat analysis will be applied to maintain the benefits of randomization and avoid introducing bias due to non-adherence or dropouts. By analyzing participants as part of their original assigned group, the ITT analysis provides a more conservative estimate of treatment effects, reflecting real-world scenarios where not everyone perfectly adheres to the assigned treatment.

Randomization:

Block randomization will be used to determine which side of teeth (right or left side quadrants) the bulk-fill composite will be used to bond the brackets in each participant. This will be controlled by a research faculty member of the Section of Dentistry assigned to the research by the Clinical Trials Unit AKUH.

Random Sequence Generation:

In this two-armed study, fifteen blocks each with a block size of four with any of the following six-possible allocation sequences for two treatment arms will be generated.

(1) AABB, (2) BBAA, (3) ABAB, (4) BABA, (5) ABBA, (6) BAAB The blocks to be utilized and their order will be determined by the research Faculty member using sealed envelopeTM online software.

Allocation Sequence Concealment:

The treatment allocation pattern determined against each participant's ID (01-58, in ascending order) by the research faculty member, will be printed individually on paper. These papers will be sealed in an opaque envelope with the participants' ID mentioned over the envelope by a team member independent of the trial.

Enrollment:

After obtaining approval from the ERC (AKUH), each participant fulfilling the inclusion criteria for the study and consenting to participate in the trial will be assigned a participant ID.

Implementation:

During the recruitment of the participants in the trial, the sealed envelope for a participant ID will be opened to reveal the random sequence by the enrolling team member.

Blinding:

The study investigators, patients and assessors will not be blinded during the trial. The patients will be recruited by the co-principal investigator. All the measurements will be recorded by the co-investigator on the study proforma.

Inclusion Criteria:

* Patients aged between 12 - 40 years
* Patients undergoing fixed orthodontic treatment
* Patients with good oral hygiene, with grade 1 or below on plaque and gingival indices
* All patients who will sign the informed consent/assent form

Exclusion Criteria:

* Patients with enamel surface defects
* Patients with any periodontal disease i.e. gingivitis or periodontitis
* Patients with any systemic diseases i.e. diabetes and hypertension
* Pregnant or nursing females
* Patients with craniofacial syndromes
* Subjects with a previous history of orthodontic or orthopedic treatment

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged between 13 - 40 years

  * Patients undergoing fixed orthodontic treatment
  * Patients with good oral hygiene, with grade 1 or below on plaque and gingival indices
  * All patients who will sign the informed consent/assent form

Exclusion Criteria:

* • Patients with enamel surface defects

  * Patients with any periodontal disease i.e. gingivitis or periodontitis
  * Patients with any systemic diseases i.e. diabetes and hypertension
  * Pregnant or nursing females
  * Patients with craniofacial syndromes
  * Subjects with a previous history of orthodontic or orthopedic treatment

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival Time of Orthodontic Bracket Bond | First, at the time of brackets bonding (T0), after one month (T1), two months (T2) and three months follwow-up (T3).
  The number of days the bonded orthodontic brackets remain adhered to the tooth surface without failure. Bracket bond failure will be recorded at each follow-up visit, and survival time will be calculated for each bracket in both intervention groups (bulk fill composite vs conventional composite). The aim is to compare the average survival duration between the two materials over the study period.

SECONDARY OUTCOMES:
Plaque Accumulation and Gingival Health | First, at the time of brackets bonding (T0), after one month (T1), two months (T2) and three months follwow-up (T3).
  Dental plaque accumulation and gingival health will be assessed using the Plaque Index and Gingival Index, respectively. These clinical indices will be measured around brackets bonded with bulk fill composite and conventional composite. The comparison will help evaluate whether the type of bonding material influences oral hygiene status and gingival inflammation during fixed orthodontic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT07155343/Prot_SAP_000.pdf
  • Informed Consent Form: Adults informed consent form (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT07155343/ICF_001.pdf
  • Informed Consent Form: Parental informed consent form (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT07155343/ICF_002.pdf
  • Informed Consent Form: Adolescent informed consent form (2024-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT07155343/ICF_003.pdf